CLINICAL TRIAL: NCT01846390
Title: A Phase I Study of Romidepsin, Gemcitabine, Dexamethasone and Cisplatin Combination Therapy in the Treatment of Peripheral T-Cell and Diffuse Large B-Cell Lymphoma
Brief Title: Romidepsin, Gemcitabine, Dexamethasone and Cisplatin in the Treatment of Peripheral T-Cell and Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY15
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2019-11

CONDITIONS: Peripheral T-Cell Lymphoma; Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Large B-Cell, Diffuse | interventions — Gemcitabine; Dexamethasone; Cisplatin; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- romidepsin, gemcitabine, dexamethasone and cisplatin (Experimental): A traditional phase I dose escalation design is proposed to assess the feasibility and tolerability of romidepsin in combination with GDP, where treatment will be escalated. Treatment will be given for 6 cycles unless there is evidence of progression prior to completion of the 6 cycles or tolerability to the regimen is not sustained.
  Interventions: Drug: Gemcitabine; Drug: Dexamethasone; Drug: Cisplatin; Drug: Romidepsin

INTERVENTIONS:
Drug: Gemcitabine — Group 1 = 1000 mg/m2 D1, D8. Subsequent dose levels according to toxicity = 600-1000 mg/m2 D1, D15.
Drug: Dexamethasone — 40 mg D1 - D4
Drug: Cisplatin — 75 mg/m2 D1
Drug: Romidepsin — Dose Level 0 - 6 mg/m2 D1, D8. Subsequent dose levels according to toxicity 6-14 mg/m2 D1, D15.

SUMMARY:
This research is being done because it is not yet known what dose of romidepsin in combination with gemcitabine, dexamethasone, and cisplatin (GDP) can be given safely to patients with peripheral T-cell lymphoma, nor what type and severity of side effects will result from the combination of these treatments. This research is also being done because it is not clear if the addition of the new drug romidepsin to treatment with GDP can offer better results and longer survival.

DETAILED DESCRIPTION:
The purpose of this study is to find the highest dose of romidepsin that can safely be given in combination with gemcitabine, dexamethasone, and cisplatin (GDP) without causing very severe side effects that are not tolerable. This is done by starting at a dose lower than the one that does not cause side effects in animals. Patients are given romidepsin and GDP and watched very closely to see what side effects they have and to make sure the side effects are not severe. If the side effects are not severe, then more patients are asked to join the study and are given a higher dose of romidepsin (with GDP). Patients joining the study later on will get higher doses of romidepsin (with GDP) than patients who join earlier. This will continue until a dose is found that causes severe but temporary side effects. Doses higher than that will not be given.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed PTCL. Biopsy proof of disease at initial diagnosis is mandatory. A biopsy at relapse is preferred but not mandatory.
* Patients must have received one or two previous regimens of therapy for their disease (salvage chemotherapy plus autologous stem cell transplantation is considered to be one regimen).
* Clinically and / or radiologically measurable disease (1 site bidimensionally measurable). Measurements / evaluations must be done within 28 days prior to registration.
* Age 18 to 75 years.
* ECOG performance status 0, 1 or 2.
* Life expectancy of ≥ 90 days (3 months).
* Laboratory Requirements: (must be done within 7 days of registration)

Hematology:

* Granulocytes (AGC) ≥ 1.0 x 10^9/L
* Platelets ≥ 75 x 10^9/L (≥ 50 if bone marrow involvement by lymphoma)

Biochemistry:

* AST and ALT ≤ 2.5x ULN (≤ 5x ULN if hepatic involvement of disease)
* Serum total bilirubin ≤ 1.5x ULN (≤ 3x ULN if hepatic involvement of disease, or ≤5x ULN if Gilberts Disease)
* Serum Potassium ≥ 3.8 mmol/L*
* Serum Magnesium ≥ 0.85 mmol/L* * NB: Patients with potassium and magnesium levels below these values are eligible if supplementation has corrected these deficits. This supplementation should continue throughout the course of the study.

  * Calculated creatinine clearance (Cockcroft-Gault formula) of ≥ 50 mL /min.
  * Women must be post-menopausal, surgically sterile or use reliable forms of contraception while on study and for 90 days after discontinuing therapy. Women of childbearing potential must have a pregnancy test taken and proven negative within 7 days prior to registration and must not be lactating.
  * Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements.
  * Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial.
  * In accordance with NCIC CTG policy, protocol treatment is to begin within 2 working days of patient registration.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer and superficial bladder cancer, curatively treated in-situ cancer of the cervix or breast or localized excised prostate cancer, or other solid tumours curatively treated with no evidence of disease for ≥ 3 years.
* Central nervous system involvement, meningeal or parenchymal. Patients with CNS disease at initial presentation and who are in a CNS CR at the time of relapse are eligible. MRI scanning and / or lumbar puncture should be performed if there is clinical suspicion of active CNS disease.
* HIV, active hepatitis B or current hepatitis C infection. (Hepatitis B core antibody positive, surface antigen negative patients allowed if concurrent anti-viral prophylaxis is administered. Patients with a past history of hepatitis C who have eradicated the virus are eligible.)
* Any serious active disease or co-morbid medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from participating (according to investigator's decision).
* Patients with serious cardiac illness or condition including, but not limited to:

  * history of documented congestive heart failure (CHF)
  * systolic dysfunction (LVEF < 45% by MUGA or ECHO)
  * high risk uncontrolled arrhythmias (ventricular tachycardia, high-grade AV-block, supraventricular arrhythmias which are not adequately rate-controlled)
  * unstable angina pectoris requiring anti-anginal medication
  * clinically significant valvular heart disease
  * evidence of transmural infarction on ECG
  * New York Heart Association (NYHA) Class III or IV functional status
  * patients with congenital long QT syndrome, history of significant cardiovascular disease and/or taking drugs leading to significant QT prolongation
  * patients with QTc > 480 msec are not eligible
* Pregnant or lactating females or women of childbearing potential not willing to use an adequate method of birth control for the duration of the study.
* Patients with active or uncontrolled infections, or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol are not eligible.
* Patients are not eligible if they have a known hypersensitivity to the study drugs or their components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of combined romidepsin, gemcitabine, dexamethasone and cisplatin. | 48 months
  Combination of GDP with romidepsin at the maximum tolerated doses of these agents will identify the combination regimen for comparison in the subsequent randomized phase II trial; if romidepsin appears to improve the activity of GDP, then this will move forward to a formal phase III comparison to CHOP.
  Primary end points are toxicity, the maximum administered dose and the recommended phase II dose.

SECONDARY OUTCOMES:
Number of patients with adverse events | 48 months
  Adverse events by grade, dose level and total incidence; vital signs will be summarized and DLTs reported separately

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Reiman, Study Chair — Atlantic Health Sciences Corp - Saint John Regional Hospital, Saint John NB Canada; Kerry J Savage, Study Chair — BCCA Vancouver Cancer Centre, Vancouver BC Canada
Locations (6):
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Regional Health Authority B, Zone 2, Saint John, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Result] Reiman T, Savage KJ, Crump M, Cheung MC, MacDonald D, Buckstein R, Couban S, Piliotis E, Imrie K, Spaner D, Shivakumar S, Kuruvilla J, Villa D, Shepherd LE, Skamene T, Winch C, Chen BE, Hay AE. A phase I study of romidepsin, gemcitabine, dexamethasone and cisplatin combination therapy in the treatment of peripheral T-cell and diffuse large B-cell lymphoma; the Canadian cancer trials group LY.15 studydagger. Leuk Lymphoma. 2019 Apr;60(4):912-919. doi: 10.1080/10428194.2018.1515937. Epub 2018 Oct 10. PMID 30301414